CLINICAL TRIAL: NCT03985514
Title: Optimized Treatment for Uncomplicated Acute Appendicitis; Active Observation With or Without Antibiotic Treatment
Brief Title: Acute Appendicitis: Active Observation With and Without Antibiotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: App 2018
Record Dates: First submitted 2018-11-09; First posted 2019-06-13 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Piperacillin; Tazobactam; Piperacillin, Tazobactam Drug Combination; Ciprofloxacin; Metronidazole

STUDY DESIGN:
Intervention Model Description: Selected patients with assumed uncomplicated acute appendicitis are allocated to groups "Active observation" or "Antibiotic treatment" in a 1:1 ratio.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic treatment (Active Comparator): Patients will receive in-hospital intravenous antibiotics (Piperacillin/Tazobactam, 4 gram x 3), followed by 8-10 days of out-hospital oral antibiotic treatment (Ciprofloxacin 500 mgx2,Flagyl 400 mgx3). Surgery if no symptom relif occur.
  Interventions: Drug: Antibiotic treatment (Piperacillin/Tazobactam, 4 gram x 3), followed by 8-10 days of out-hospital oral antibiotic treatment (Ciprofloxacin 500 mgx2,Flagyl 400 mgx3).
- Clinical observation (Other): Patients are followed by in-hospital "Active observation" (watchful waiting) according to clinical routine. Patients are observed until either, recovery and dismissal from hospital, or decision for intervention (surgery) is taken.
  Interventions: Other: Active observation

INTERVENTIONS:
Drug: Antibiotic treatment (Piperacillin/Tazobactam, 4 gram x 3), followed by 8-10 days of out-hospital oral antibiotic treatment (Ciprofloxacin 500 mgx2,Flagyl 400 mgx3). — Intravenous antibiotic treatment x 3, followed by oral antibiotics for 8-10 Days.
  Other Names: Piperacillin/Tazobactam; Ciprofloxacin; Flagyl
  Arms: Antibiotic treatment
Other: Active observation — In-hospital observation without antibiotics
  Arms: Clinical observation

SUMMARY:
This study evaluates if early provision of antibiotics is a superior treatment compared to "traditional wait and see" with regard to symptom relief for suspected acute uncomplicated appendicitis.

DETAILED DESCRIPTION:
Recent long-term follow up results of antibiotic treatment of acute appendicitis in unselected populations indicate that approximately 70-80 % of patients respond to antibiotics, while the remaining 20-25% need an operation. Antibiotic treatment was associated with significantly fewer severe and non-severe complications compared to surgery. Therefore, antibiotic treatment can be regarded as safe and effective initial treatment of acute appendicitis based on evidence.

However, it remains to be evaluated to what extent antibiotic treatment is more effective compared to the most conservative application of procedures in the care of patients with acute appendicitis. A well- recognized approach in Sweden is watchful waiting at in-hospital conditions. A certain number of patients with suspected uncomplicated appendicitis will likely recover without any active treatment, but controlled evidence are lacking to what extent such recoveries may occur in the short- and long-term perspective.

The hypothesis is that antibiotic treatment is superior to active observation with regard to symptom relief at suspected acute appendicitis in selected patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected appendicitis.
* Age<60 years.
* C-reactive protein < 60 mg/L.
* White blod cell Count (leucocytes) < 13 e9 /L.

Exclusion criteria:

* Pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with no symptom relief | 48 hours
  No symptom relief and surgery is deemed necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Lundholm, Professor, Principal Investigator — Göteborg University
Locations (1):
- Department of surgery, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No